CLINICAL TRIAL: NCT03245658
Title: The Effect of Medical Cannabis Inpatients With Palliative Pancreatic Cancer
Brief Title: The Effect of Cannabis in Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Organization was changed. The staff was relocated.
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-17000277
Record Dates: First submitted 2017-03-21; First posted 2017-08-10 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Neoplasms Pancreatic; Cachexia; Cancer; Cannabis; Appetite Loss; Palliative Medicine; Morbidity; Mortality
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia; Neoplasms; Marijuana Abuse; Anorexia | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THC and CBD Mixture (Experimental): 32 patients with palliative pancreatic cancer, intervention with oral drops of THC, 25mg/ml and CBD 50mg/ml, daily administered for 4 weeks
  Interventions: Drug: THC and CBD Mixture
- Control (No Intervention): 32 patients with palliative pancreatic cancer, no experimental treatment,

INTERVENTIONS:
Drug: THC and CBD Mixture — Individually titrated doses on daily basis
  Other Names: Medical cannabis oral drops
  Arms: THC and CBD Mixture

SUMMARY:
Cannabinoids are known to increase appetite, but THC components have psychogenic properties too. CBD is the main component in the plant, and have only minimal psychogenic effects. The aim was to test the appetite stimulating effects of CBD in patients with pancreatic cancer in palliative treatment.

DETAILED DESCRIPTION:
Randomization of consecutive patients who wanted to participate to a daily dose of CBD or not as a supplement to the standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult, palliative pancreatic cancer diagnosis, weight loss > 5%, understand and read Danish.

Exclusion Criteria:

* Regular use of cannabis, psychiatric disorders, alcohol abuse, life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-06 (Estimated); Primary Completion 2018-05-06 (Estimated); Study Completion 2018-10-06 (Estimated)

PRIMARY OUTCOMES:
Energy and protein intake | The outcome measure will be assessed at day 0 and at week 4
  Dietary history (% of estimated needs - NRS 2002)

SECONDARY OUTCOMES:
Lean body mass | The outcome measure will be assessed at day 0 and at week 4
  Bioimpedance (% of body weight, kg)
Appetite 1 | The outcome measure will be assessed at day 0 and at week 4
  VAS (cm on 10 cm scale)
Appetite 2 | The outcome measure will be assessed at day 0 and at week 4
  Dietary history (VAS (cm on 10 cm scale))
Appetite 3 | The outcome measure will be assessed at day 0 and at week 4
  EORTC QLQ-C30 (score, standard for the Quality of Life entity)
Appetite 4 | The outcome measure will be assessed at day 0 and at week 4
  EORTC QLQ-PAN26 (score, standard for the Quality of Life entity)
Quality of life 1 | The outcome measure will be assessed at day 0 and at week 4
  EORTC QLQ-C30 (score, standard for the Quality of Life entity)
Quality of life 2 | The outcome measure will be assessed at day 0 and at week 4
  EORTC QLQ-PAN26 (score, standard for the Quality of Life entity)
Quality of life 3 | The outcome measure will be assessed at day 0 and at week 4
  VAS (VAS (cm on 10 cm scale))
Pain 1 | The outcome measure will be assessed at day 0 and at week 4
  EORTC QLQ-C30 (score, standard for the Quality of Life entity)
Pain 2 | The outcome measure will be assessed at day 0 and at week 4
  EORTC QLQ-PAN26 (score, standard for the Quality of Life entity)
Pain 3 | The outcome measure will be assessed at day 0 and at week 4
  VAS (VAS (cm on 10 cm scale))
Mortality (8 weeks) | 8 weeks
  Patient records, national register

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, MPA, Principal Investigator — University of Copenhagen
Locations (1):
- Department of clinical oncology, Næstved-Roskilde Hospital, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perras C. Sativex for the management of multiple sclerosis symptoms. Issues Emerg Health Technol. 2005 Sep;(72):1-4. PMID 16317825
- [Result] Gartner S, Kruger J, Aghdassi AA, Steveling A, Simon P, Lerch MM, Mayerle J. Nutrition in Pancreatic Cancer: A Review. Gastrointest Tumors. 2016 May;2(4):195-202. doi: 10.1159/000442873. Epub 2016 Jan 8. PMID 27403414
- [Result] Ware MA, Daeninck P, Maida V. A review of nabilone in the treatment of chemotherapy-induced nausea and vomiting. Ther Clin Risk Manag. 2008 Feb;4(1):99-107. doi: 10.2147/tcrm.s1132. PMID 18728826
- [Result] Grotenhermen F. Pharmacokinetics and pharmacodynamics of cannabinoids. Clin Pharmacokinet. 2003;42(4):327-60. doi: 10.2165/00003088-200342040-00003. PMID 12648025
- [Result] Slatkin NE. Cannabinoids in the treatment of chemotherapy-induced nausea and vomiting: beyond prevention of acute emesis. J Support Oncol. 2007 May;5(5 Suppl 3):1-9. PMID 17566383
- [Result] Johnson JR, Lossignol D, Burnell-Nugent M, Fallon MT. An open-label extension study to investigate the long-term safety and tolerability of THC/CBD oromucosal spray and oromucosal THC spray in patients with terminal cancer-related pain refractory to strong opioid analgesics. J Pain Symptom Manage. 2013 Aug;46(2):207-18. doi: 10.1016/j.jpainsymman.2012.07.014. Epub 2012 Nov 8. PMID 23141881
- [Result] Johnson JR, Burnell-Nugent M, Lossignol D, Ganae-Motan ED, Potts R, Fallon MT. Multicenter, double-blind, randomized, placebo-controlled, parallel-group study of the efficacy, safety, and tolerability of THC:CBD extract and THC extract in patients with intractable cancer-related pain. J Pain Symptom Manage. 2010 Feb;39(2):167-79. doi: 10.1016/j.jpainsymman.2009.06.008. Epub 2009 Nov 5. PMID 19896326
- [Result] Reuter SE, Martin JH. Pharmacokinetics of Cannabis in Cancer Cachexia-Anorexia Syndrome. Clin Pharmacokinet. 2016 Jul;55(7):807-812. doi: 10.1007/s40262-015-0363-2. PMID 26883879
- [Result] Gamage TF, Lichtman AH. The endocannabinoid system: role in energy regulation. Pediatr Blood Cancer. 2012 Jan;58(1):144-8. doi: 10.1002/pbc.23367. PMID 22076835
- [Result] Fox KM, Brooks JM, Gandra SR, Markus R, Chiou CF. Estimation of Cachexia among Cancer Patients Based on Four Definitions. J Oncol. 2009;2009:693458. doi: 10.1155/2009/693458. Epub 2009 Jul 1. PMID 19587829
- [Result] Gullett N, Rossi P, Kucuk O, Johnstone PA. Cancer-induced cachexia: a guide for the oncologist. J Soc Integr Oncol. 2009 Fall;7(4):155-69. PMID 19883531
- [Result] Blum D, Omlin A, Fearon K, Baracos V, Radbruch L, Kaasa S, Strasser F; European Palliative Care Research Collaborative. Evolving classification systems for cancer cachexia: ready for clinical practice? Support Care Cancer. 2010 Mar;18(3):273-9. doi: 10.1007/s00520-009-0800-6. PMID 20076976
- See also: review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4924449/